CLINICAL TRIAL: NCT00006421
Title: Breast Imaging Screening Studies in Women at High Genetic Risk of Breast Cancer: Annual Follow-up Study
Brief Title: Breast Imaging Studies in Women at High Genetic Risk of Breast Cancer: Annual Follow-Up Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010009; 01-C-0009; NCT00012415 (obsolete NCT alias)
Record Dates: First submitted 2000-10-27; First posted 2000-10-30 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-06-26

CONDITIONS: Breast Cancer
Keywords: Breast MRI; Nipple Aspirate Fluid; Transvaginal ultrasound; Ductal lavage
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: 2-Fluorodeoxyglucose

SUMMARY:
This study will explore new screening methods for early detection of breast and ovarian cancer in women at high risk for these diseases, because they have an altered breast cancer 1 (BRCA1) or breast cancer 2 (BRCA2) gene. It will also try to determine if breast tissue characteristics in women with a BRCA1 or BRCA2 mutation differ from those in women with a normal gene.

Premenopausal women between 25 and 45 years of age who have participated in National Cancer Institute studies for families or individuals at high genetic risk of cancer (78-C-0039 or 99-C-0081) and who have at least a 50 percent probability of carrying an altered BRCA1 or BRCA2 gene may be eligible for this study.

At the first visit, participants will have from 4 to 24 tablespoons of blood drawn and will be interviewed about breast and ovarian cancer risk factors, family and personal history of cancer, history of pregnancies, use of oral contraceptives and other hormones and drugs, and previous surgery on the breasts and ovaries. In addition, they will undergo the following procedures:

Routine breast and ovarian cancer screening for high-risk women, including a mammogram, breast and pelvic exam, instruction in breast self-examination, CA 125 blood test and transvaginal ultrasound of the ovaries.

Magnetic Resonance Imaging (MRI) of the breast MRI uses a strong magnetic field to show structural and chemical changes in tissues.

Breast Duct Lavage In this procedure samples of fluid and cells from the lining of the breast milk ducts are collected to look for cancerous or pre-cancerous cell changes.

Positron Emission Tomography (PET) scan PET scanning will be done only in participants whose mammogram or MRI findings require additional evaluation. This diagnostic test is based on differences in how cells take up and use glucose (sugar), one of the body s main fuels.

Annual follow-up visits will be scheduled for 3 years and will include routine high-risk screening as described above, blood draw, update of family history and risk factors, breast MRI, breast duct lavage and, if there are changes on the MRI or mammogram that need further evaluation, the PET will be repeated.

DETAILED DESCRIPTION:
Background:

* Women who carry mutations in genes such as BRCA1/2 have a higher lifetime risk of breast cancer (BC) and are at risk of developing BC at earlier ages than women in the general population.
* Prophylactic mastectomy and/or oophorectomy may be used to decrease risk and intensified mammographic and magnetic resonance imaging (MRI) surveillance may allow earlier diagnosis; however, prophylactic mastectomy has not been shown to convey survival advantage over more conservative management.
* Greater breast tissue density and low BC incidence result in a lower positive predictive value of mammography in premenopausal women as compared to postmenopausal women (PPV=0.04 for women aged 40-49).
* This study explores whether high-risk breast imaging phenotypes may be identified by comparing imaging characteristics of mutation carriers/non-carriers using two imaging modalities: mammography and MRI.
* Nipple Aspiration Fluid collection (NAF) and breast duct lavage will be used to obtain cytologic materials which may be used as an adjunct to breast imaging for the early detection of epithelial atypia and pre-invasive cancer.

Objectives:

* Compare four outcomes including two mammographic density measures (qualitative and semiquantitative), fibroglandular volume measure using MRI, and contrast enhancement measure using MRI (both semiquantitative) in mutation carriers/non-carriers to improve lesion detection
* Explore non-ionizing approaches (MRI) to BC screening because the effects of ionizing radiation due to mammography are unknown.
* Use NAF and/or BDL to obtain epithelial cell samples and correlate cytologic and imaging findings.
* Gather prospective data on the transformation from normal/hyperplastic/pre-invasive/invasive disease in BRCA1/2 mutation carriers/non-carriers through molecular/genetic studies of breast tissue (via biopsy of radiographic abnormalities) or breast fluid (via BDL and/or nipple aspiration) and develop molecular markers for early detection of epithelial atypia/pre-invasive cancer.
* Assess the psychosocial impact of participation in a BC screening program.

Eligibility:

* Women 25-56 years of age carrying a known BRCA1/2 deleterious mutation.
* Women between the ages of 25 -56 who are first- or second- degree relatives of individuals with a deleterious BRCA1/2 mutation.
* Women aged 25-56 who are first- or second- degree relatives of individuals with BRCA-associated cancers in families with documented BRCA mutations.

Design:

* Prospective cohort study of 200 women to gather data on the evolution of epithelial cell/molecular changes in BRCA1/2 mutation carriers, by collecting/analyzing NAF, BDL fluid, biopsy tissues (when indicated), and serum/lymphocytes; samples are stored for future studies.
* Women complete questionnaires and undergo breast/pelvis examination, transvaginal ultrasonography, serum pregnancy test, fasting glucose, electrolytes, BUN, creatinine and CA 125. Standard four view mammogram and breast MRI are performed on study entry and annually for three additional years.

ELIGIBILITY:
* INCLUSION CRITERIA - Annual Follow-up Study:

To participate in the Annual Follow-up Study, a woman must:

Be at least 25 years of age (or 5 years younger than the age at diagnosis of the youngest family member with a tumor associated with the Breast-Ovarian Cancer Syndrome) and less than 56 years of age.

Must be:

A known BRCA1 or BRCA2 deleterious mutation carrier

OR

A first- or second- degree relative of an individual known to carry a deleterious BRCA1 or BRCA2 mutation

OR

A first- or second- degree relative of an individual with a tumor associated with the Breast-Ovarian Cancer Syndrome in a family with a known BRCA mutation.

Have undergone genetic counseling and risk assessment.

Agree to release of genetic test result for stratification purposes, whether or not she has chosen to receive individual test results for clinical decision-making.

Have an ECOG performance status of 0-1.

Be able to provide informed consent.

Have at least one non-irradiated breast.

EXCLUSION CRITERIA - Annual Follow-up Study:

Any of the following will result in exclusion from the Annual Follow-up Study:

Pregnancy or lactation within 6 months of enrollment.

Abnormal CA-125 level.

Bilateral breast cancer, ovarian (any stage) or breast cancer (Stage IIB or worse) unless relapse free for 5 years prior to the time of enrollment.

Patients with DCIS, Stage I and Stage II breast cancer are eligible provided that it has been at least 6 months from the completion of primary therapy (surgery, radiation, and chemotherapy as applicable). Tamoxifen and aromatase inhibitor adjuvant therapy is allowed.

Patients with DCIS, Stage I and Stage II breast cancer who have had a local relapse after primary treatment are not eligible unless they have been relapse free for 5 years prior to the time of enrollment.

History of other invasive cancer unless relapse free for 5 years prior to the time of enrollment. Non-Melanoma skin cancer or cervical carcinoma in situ are excepted.

Previous bilateral mastectomy or bilateral radiation therapy.

Weigh over 136 kilograms.

Allergy to gadolinium.

Allergy to lidocaine or Marcaine (bupivacaine). (excluded from breast duct lavage only).

Subareolar or other surgery of the breast to be studied which might disrupt the ductal systems. For example, papilloma resection, biopsy or fine needle aspirations (FNAs) within 2 cm of the nipple might disrupt the ductal systems. Biopsies or FNAs greater than 2 cm from the nipple are acceptable. (Excluded from ductal lavage only)

A breast implant or prior silicone injections in the breast to be studied. (Exclude from breast ductal lavage only)

Active infections or inflammation in a breast to be studied. (breast ductal lavage only)

Medical or psychiatric disorder which, in the opinion of the Principal Investigator, would preclude informed consent or ability to participate in clinical research.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study explores whether high-risk breast imaging phenotypes may be identified by comparing imaging characteristics of mutation carriers /non-carriers using two imaging modalities: mammography and MRI. This is a prospective cohort study of 200 women to gather data on the evolution of epithelial cell/molecular changes in BRCA1/2 mutation carriers, by collecting/analyzing NAF, BDL fluid, biopsy tissues (when indicated), and serum/lymphocytes; samples are stored for future studies. Eligible study participants include: 1)Women 25-56 years of age carrying a known deleterious mutation; 2) BRCA1/2@@@Women between the ages of 25 56 who are first- or second- degree relatives of individuals with a deleterious mutation. BRCA1/2, and 3)Women aged 25-56 who are first- or second- degree relatives of individuals with associated cancers in families with documented BRCA- BRCA mutations.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2000-10-25 (Actual)

PRIMARY OUTCOMES:
Differences in measures of mammographic density and MRI fibroglandular volume between mutation positive and mutation negative women | 1/1/2001-12/31/2011
  Compare four outcomes including two mammographic density measures (qualitative and semi-quantitative), fibroglandular volume measure using MRI, and contrast enhancement measure using MRI (both semiquantitative) in mutation carriers/non-carriers to improve lesion detection
Cytologic cell counts, mammographic density and MRI fibroglandular volume | 1/1/2001-12/31/2011
  Use NAF and/or BDL to obtain epithelial cell samples and correlate cytologic and imaging findings.
Obtain biologic materials in participants who undergo clinically indicated surgical procedures and NAF/BDL over time and correlate with outcomes of breast screening. | 1/1/2001-12/31/2011
  Gather prospective data on the transformation from normal/hyperplastic/pre-invasive/invasive disease in BRCA1/2 mutation carriers/non-carriers through molecular/genetic studies of breast tissue (via biopsy of radiographic abnormalities) or breast fluid (via BDL and/or nipple aspiration) and develop molecular markers for early detection of epithelial atypia/pre-invasive cancer.
Use questionnaires and interviews to evaluate the impact, emotional outcomes and decision-making in study participants | Study period
  Assess the psychosocial impact of participation in a BC screening program.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Savage, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Koehly LM, Peters JA, Kenen R, Hoskins LM, Ersig AL, Kuhn NR, Loud JT, Greene MH. Characteristics of health information gatherers, disseminators, and blockers within families at risk of hereditary cancer: implications for family health communication interventions. Am J Public Health. 2009 Dec;99(12):2203-9. doi: 10.2105/AJPH.2008.154096. Epub 2009 Oct 15. PMID 19833996
- [Background] Loud JT, Thiebaut AC, Abati AD, Filie AC, Nichols K, Danforth D, Giusti R, Prindiville SA, Greene MH. Ductal lavage in women from BRCA1/2 families: is there a future for ductal lavage in women at increased genetic risk of breast cancer? Cancer Epidemiol Biomarkers Prev. 2009 Apr;18(4):1243-51. doi: 10.1158/1055-9965.EPI-08-0795. Epub 2009 Mar 31. PMID 19336560
- [Background] Gierach GL, Loud JT, Chow CK, Prindiville SA, Eng-Wong J, Soballe PW, Giambartolomei C, Mai PL, Galbo CE, Nichols K, Calzone KA, Vachon C, Gail MH, Greene MH. Mammographic density does not differ between unaffected BRCA1/2 mutation carriers and women at low-to-average risk of breast cancer. Breast Cancer Res Treat. 2010 Aug;123(1):245-55. doi: 10.1007/s10549-010-0749-7. Epub 2010 Feb 4. PMID 20130984
- [Derived] Ersig AL, Werner-Lin A, Hoskins L, Young J, Loud JT, Peters J, Greene MH. Legacies and Relationships: Diverse Social Networks and BRCA1/2 Risk Management Decisions and Actions. J Fam Nurs. 2019 Feb;25(1):28-53. doi: 10.1177/1074840718815844. Epub 2018 Dec 12. PMID 30537877
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-C-0009.html